CLINICAL TRIAL: NCT06226012
Title: Effect of Pulsed Magnetic Field Versus Low Level Laser Therapy on Functional Performance in Children With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shrouk Abd Elmohsen Taha Basiony Elnhrawy (Other)
Responsible Party: Sponsor-Investigator, Shrouk Abd Elmohsen Taha Basiony Elnhrawy, bachelors degree of physical therapy, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EG,KFS lab Research 00
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group (A) received Pulsed magnetic field therapy in addition to traditional exercise program
  Interventions: Device: pulsed magnetic field
- Group B (Experimental): Group (B) received Low level laser therapy in addition to traditional exercise program
  Interventions: Device: Low level laser

INTERVENTIONS:
Device: pulsed magnetic field — Children in this group received pulsed magnetic therapy in addition to traditional exercise program
  Arms: Group A
Device: Low level laser — Children in this group received low level laser therapy in addition to traditional exercise program
  Arms: Group B

SUMMARY:
the purpose of this study is to compare between the effect of pulsed magnetic field versus low level laser therapy on functional performance in children with juvenile idiopathic arthritis

DETAILED DESCRIPTION:
This study directed to investigate effect of pulsed magnetic field versus low level laser therapy on functional performance in children with juvenile idiopathic arthritis children with juvenile idiopathic arthritis suffer from some problems such as pain, swelling and limited motion in knee joints here in this study i used these devices to help in solving these problems pain was measured by visual analogue scale swelling was measured by tape measurement and Range of motion was measured by digital geniometre

ELIGIBILITY:
Inclusion Criteria:

* 1 Confirmed diagnosis of Juvenile Idiopathic Arthritis (JIA).
* 2 Polyarticular onset of JIA with bilateral involvement of the knee joint.
* 3 Age between 8 and 16 years
* 4 Stable conditions (i.e., receive stable doses of medications in the past three months).
* 5 Not participating in a regular exercise program in the past six months.

Exclusion Criteria:

* 1 Fixed deformities
* 2 History of joint surgery
* 3 Ankylosing or fractures
* 4 Bone destruction ( erosive changes of the knee joints ).

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Swelling | 3 months
  We used Tape Measurement to measure Swelling
Sensation of Pain | 3 months
  we used Visual Analogue Scale (VAS) to measure pain. the scale ranged from 0 to 10. ( 0 means no pain and 10 means maximum pain
Range of motion | 3 months
  we used digital geniometer to measure range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Kafr Elsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided